CLINICAL TRIAL: NCT06236971
Title: Effect of Lateral Positions on the Shape of Upper Airway Under Sedation
Brief Title: Effect of Lateral Positions on the Shape of Upper Airway
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Zhejiang Provincial Tongde Hospital (Other)
Responsible Party: Principal Investigator, xiangming fang, Director, Head of Anesthesiology and Critical Care, Principal Investigator, Professor, First Affiliated Hospital of Zhejiang University
Other Study IDs: airway
Record Dates: First submitted 2024-01-13; First posted 2024-02-01 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Airway Remodeling; Radiography in Otolaryngology; Position; Patency; Morphology
MeSH Terms: conditions — Airway Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI scanning: The subjects are receiving MRI scanning first in the supine position, and then in the lateral position. The field of view was determined from the length and girth of each patient's head, at least including the skull base to the level of tracheal bifurcation.
  Interventions: Behavioral: MRI scanning first at supine position and then turn into lateral position

INTERVENTIONS:
Behavioral: MRI scanning first at supine position and then turn into lateral position — Magnetic resonance imaging was used to scan the upper airway of sedated subjects, first at supine position and then turn into lateral position.

SUMMARY:
The severity and frequency of respiratory events is increased in the supine body posture compared with the lateral position in emergency, difficult airway patients. The mechanism responsible is not clear but may relate to the effect of position on upper airway shape and size. 3D finite element model of upper airway filling based on MRI image reconstruction can effectively reflect the anatomy of the upper airway. This study compared the effect of body position on upper airway shape and size in individuals with lateral position among sedated subjects.

DETAILED DESCRIPTION:
Anesthesiologists may encounter situations in which a accidental loss of airway patency occurs in patients in a lateral patient position during surgery. Intubation is required in the lateral position in cases of oropharyngeal bleeding to reduce the risk of aspiration, or in airway management in some patients with limited posture. The severity and frequency of respiratory events is increased in the supine body posture compared with the lateral position in emergency, difficult airway patients. The mechanism responsible is not clear but may relate to the effect of position on upper airway shape and size secondary to gravitational effects. Lateral positioning decreases upper airway obstruction in sleeping individuals, children breathing spontaneously, and adults during general anesthesia. The mechanical upper airway properties may become the dominant factor governing upper airway collapsibility during sedation due to the significant depression of consciousness and the impairment of neural mechanisms controlling compensatory neuromuscular responses. Anesthesiologists and surgeons who are responsible for airway management during procedures under sedation and the perioperative period should be well versed with the physiological and pathophysiological mechanisms affecting upper airway patency. 3D finite element model of upper airway filling based on MRI image reconstruction can effectively reflect the anatomy of the upper airway.

The primary aim of this study was to determine the changes in upper airway shape and size that occur when sedated, spontaneously breathing adults are placed in the lateral position. These findings may provide new guidance for the evaluation and prediction of difficult airway during clinical anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged over than 18 years and less than 100 years
2. The American Society of Anesthesiologists (ASA) score was grade I to II
3. There was no serious cardiopulmonary disease

Exclusion Criteria:

1. Unable to maintain oxygenation before or during the examination and requiring intervention
2. Those with preoperative arrhythmia requiring intervention
3. Thosewith severe hematological diseases, severe metabolic diseases, severe liver and kidney organ insufficiency
4. Those do not consent to participate in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects aged over 18 years old, ASA 1~II without serious cardiopulmonary disease, scheduled for magnetic resonance imaging scan in the supine position and followed lateral position at a tertiary hospital from January 2024 to February 2024 were enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
minimum cross-sectional area (MCSA) | through study completion, an average of 2 months
  minimum cross-sectional area (MCSA) of upper airway-related sagittal, cross-sectional, and coronal planes
minimum anteroposterior | through study completion, an average of 2 months
  minimum anteroposterior diameters
lateral diameters | through study completion, an average of 2 months
  lateral diameters
pharyngeal volume | through study completion, an average of 2 months
  pharyngeal volume

SECONDARY OUTCOMES:
three-dimensional geometrical modeling of the upper airway | through study completion, an average of 2 months
  three-dimensional geometrical modeling of the upper airway by MATALAB software
Change of heart rates (HR) in beats per minute | before examination, immediately after examination at supine position, immediately before examination at lateral position, immediately after examination at lateral position
  compared the change of HR in beats per minute between different position
Change of oxygenation (SpO2, %) | before examination, immediately after examination at supine position, immediately before examination at lateral position, immediately after examination at lateral position
  compared the change of SpO2 (%)
Change of respiratory rates (RR) in respirations per minute | before examination, immediately after examination at supine position, immediately before examination at lateral position, immediately after examination at lateral position
  compared the change of RR in respirations per minute between different position

CONTACTS AND LOCATIONS:
Overall Officials: Xiangming Fang, M.D., Principal Investigator — The First Affiliated Hospital School of MedicineZhejiang University
Locations (1):
- Tongde Hospital of Zhejiang Province, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin CY, Chen CN, Kang KT, Hsiao TY, Lee PL, Hsu WC. Ultrasonographic Evaluation of Upper Airway Structures in Children With Obstructive Sleep Apnea. JAMA Otolaryngol Head Neck Surg. 2018 Oct 1;144(10):897-905. doi: 10.1001/jamaoto.2018.1809. PMID 30242332
- [Background] Campos LD, Trindade IEK, Trindade SHK, Pimenta LAF, Kimbell J, Drake A, Marzano-Rodrigues MN, Trindade-Suedam IK. Effects of 3D Airway Geometry on the Airflow of Adults with Cleft Lip and Palate and Obstructive Sleep Apnea: A Functional Imaging Study. Sleep Sci. 2023 Nov 22;16(4):e430-e438. doi: 10.1055/s-0043-1776868. eCollection 2023 Dec. PMID 38197022
- [Background] Chen W, Ma L, Shao J, Bi C, Xie Y, Zhao S. Morphological specificity analysis of an image-based 3D model of airway filling in a difficult airway. BMC Anesthesiol. 2022 Nov 3;22(1):336. doi: 10.1186/s12871-022-01880-6. PMID 36329383
- [Background] Martinez A, Muniz AL, Soudah E, Calvo J, Suarez AA, Cobo J, Cobo T. Physiological and geometrical effects in the upper airways with and without mandibular advance device for sleep apnea treatment. Sci Rep. 2020 Mar 24;10(1):5322. doi: 10.1038/s41598-020-61467-4. PMID 32210246
- [Background] Dollinger M, Jakubass B, Cheng H, Carter SJ, Kniesburges S, Aidoo B, Lee CH, Milstein C, Patel RR. Computational fluid dynamics of upper airway aerodynamics for exercise-induced laryngeal obstruction: A feasibility study. Laryngoscope Investig Otolaryngol. 2023 Aug 19;8(5):1294-1303. doi: 10.1002/lio2.1140. eCollection 2023 Oct. PMID 37899858
- [Background] Li H, Wang W, Lu YP, Wang Y, Chen LH, Lei LP, Fang XM. Evaluation of Endotracheal Intubation with a Flexible Fiberoptic Bronchoscope in Lateral Patient Positioning: A Prospective Randomized Controlled Trial. Chin Med J (Engl). 2016 Sep 5;129(17):2045-9. doi: 10.4103/0366-6999.189069. PMID 27569229
- [Background] Hyldmo PK, Vist GE, Feyling AC, Rognas L, Magnusson V, Sandberg M, Soreide E. Is the supine position associated with loss of airway patency in unconscious trauma patients? A systematic review and meta-analysis. Scand J Trauma Resusc Emerg Med. 2015 Jul 1;23:50. doi: 10.1186/s13049-015-0116-0. PMID 26129809
- [Background] Litman RS, Wake N, Chan LM, McDonough JM, Sin S, Mahboubi S, Arens R. Effect of lateral positioning on upper airway size and morphology in sedated children. Anesthesiology. 2005 Sep;103(3):484-8. doi: 10.1097/00000542-200509000-00009. PMID 16129971
- [Background] Litman RS, Weissend EE, Shrier DA, Ward DS. Morphologic changes in the upper airway of children during awakening from propofol administration. Anesthesiology. 2002 Mar;96(3):607-11. doi: 10.1097/00000542-200203000-00016. PMID 11873035